CLINICAL TRIAL: NCT00105937
Title: Multi-center, Open Label, Long-term Study of OraVescent Fentanyl Citrate for the Treatment of Breakthrough Pain in Opioid Tolerant Cancer Patients
Brief Title: OraVescent Fentanyl (OVF) for the Treatment of Breakthrough Pain in Opioid Tolerant Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 099-15
Record Dates: First submitted 2005-03-18; First posted 2005-03-21 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2007-05

CONDITIONS: Pain; Cancer
Keywords: Cancer; Pain
MeSH Terms: conditions — Pain; Neoplasms

INTERVENTIONS:
Drug: OraVescent fentanyl citrate

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of OraVescent fentanyl to treat breakthrough pain episodes in cancer patients who are already opioid tolerant.

DETAILED DESCRIPTION:
The objective of this study is to determine the tolerability and safety of OraVescent fentanyl when used long term to relieve breakthrough pain in opioid tolerant cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Average of 1-4 breakthrough pain episodes per day
* Opioid tolerant
* Histologically documented diagnosis of a malignant solid tumor or hematological malignancy

Exclusion Criteria:

* Primary breakthrough pain is not related to cancer in any way
* Opioid or fentanyl intolerance
* Chronic obstructive pulmonary disease (COPD) or heart disease
* Sleep apnea or active brain metastases with increased cranial pressure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-04; Study Completion 2006-11

PRIMARY OUTCOMES:
Tolerability and safety of OraVescent fentanyl when used long-term

SECONDARY OUTCOMES:
Assess the effectiveness of OraVescent fentanyl
Assess the development of incremental tolerance

CONTACTS AND LOCATIONS:
Locations (43):
- United States (43):
  - Center for Pain Management, Huntsville, Alabama
  - Outcomes Research International, Tucson, Arizona
  - Arizona Clinical Research Center, Tucson, Arizona
  - Hot Spring Pain Clinic, Hot Springs, Arkansas
  - Saint Joseph's Mercy Cancer Center, Hot Springs, Arkansas
  - Arkansas Cancer Institute, Pine Bluff, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - The Cancer Prevention and Treatment Center, Soquel, California
  - Northwestern Connecticut Oncology & Hematology Associates, Torrington, Connecticut
  - Florida Institute of Medical Research, Jacksonville, Florida
  - University of Florida Shands Cancer Center at Jacksonville, Jacksonville, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Innovative Medical Research of South Florida, Miami Shores, Florida
  - Gulf Coast Oncology Association, St. Petersburg, Florida
  - Clinical Pharmacology Services, Inc, Tampa, Florida
  - Palm Beach Research, West Palm Beach, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Southeastern Gynecologic Oncology, LLC, Atlanta, Georgia
  - North Shore Cancer Research Association, Skokie, Illinois
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Southwest Oncology Associates, Lafayette, Louisiana
  - Hematology and Oncology Specialists, New Orleans, Louisiana
  - St. Agnes Healthcare, Baltimore, Maryland
  - Huron Medical Center, Port Huron, Michigan
  - Providence Cancer Institute, Southfield, Michigan
  - Bond Clinic, Inc, Rolla, Missouri
  - HealthCare Research, LLC, St Louis, Missouri
  - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - PETC Research Group, Inc., Tulsa, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Mohamed Haq, Pasadena, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - UTHCT (ATTN: Clinical Research), Tyler, Texas
  - Hunstman Cancer Institute, Salt Lake City, Utah
  - Palliative Care and Pain Medicine, Salt Lake City, Utah
  - Great Basin Clinical Research, West Point, Utah
  - Cancer Outreach Associates, PC, Abingdon, Virginia
  - MedSource Inc, Richmond, Virginia
  - University of Wisconsin Medical School, Madison, Wisconsin